CLINICAL TRIAL: NCT04530292
Title: Evaluation of the Impact of a Home-based Intervention by a Pediatric Nurse to Prevent Diabetes Imbalance Within One Year of Its Discovery in Children Whose Parents Are in a Precarious Social Situation (PRECADIAB)
Brief Title: Home Intervention and Social Precariousness in Childhood Diabetes
Acronym: PRECADIAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CHUBX 2018/56
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Pediatric type-1 diabetes; Therapeutic education; Social precariousness
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention by a pediatric nurse at the child's home (Experimental): The pediatric nurse will visit the patient's home 3 times during the first six months of the discovery of diabetes in children. These visits will be organized during the first, fourth and sixth months after the discovery of diabetes and last about 2 hours each time. An additional visit can be organized according to the needs of families.
  The pediatric nurse will ensure the implementation of learning in terms of drug therapy (modality of insulin administration, adaptation of insulin doses) and diet, according to the knowledge acquired during the initial hospitalization. She will offer her help to the families to make a connection with the school and after-school activities of the child.
  In addition to these visits, the child and his family will come to the hospital as part of the regular medical follow-up: consultations with the pediatric diabetologist at the 3rd and 6th month and at 1 year of the discovery of diabetes.
  Interventions: Behavioral: Intervention by a pediatric nurse at the child's home
- Classic strategy (for retrospective group) (No Intervention): The child and his family benefited from a consultation with a pediatric nurse at 1 month of the discovery of T1D and had medical consultations with the pediatric diabetologist at the 3rd and 6th month and at 1 year of the discovery of diabetes. The data from this group were collected in a previous study (collection of retrospective data) for children whose parents were in a precarious social situation and whose management was traditional.

INTERVENTIONS:
Behavioral: Intervention by a pediatric nurse at the child's home — The intervention will consist of a coordinated intervention by a pediatric nurse at the child's home to support the parents in the implementation of the theoretical knowledge acquired at the hospital.
  Three home visits will be set up by a nurse during the first six months of the discovery of diabetes in the child. These visits will be organized during the first, fourth and sixth months after the discovery of diabetes and last about 2 hours each time. An additional visit may be set up according to the needs of families.
  Other Names: strategy under study ( for prospective group)
  Arms: intervention by a pediatric nurse at the child's home

SUMMARY:
A pilot study of children whose families are in a precarious situation, who will benefit from a targeted at-home intervention by a pediatric nurse. Visits will be organized during the first, fourth and sixth months after the discovery of diabetes. The HbA1C measured 12 months after the diabetes diagnosis will be compared to the HbA1C obtained in an historical cohort that did not receive at-home therapeutic education.

DETAILED DESCRIPTION:
The EPICES score is an individual indicator of precariousness associated with indicators of access to health care and indicators of health. For this score, 30 is considered as the precariousness threshold. It is collected during the follow-up of our cohort of diabetic children and the data is obtained from the parent accompanying the child.

In 2016, we found in this cohort that a context of precariousness was associated with a very poor result of glycated hemoglobin (HbA1C) (Lamaraud J et al., 2017). The imbalance of diabetes was detectable as early as one year after diagnosis and persisted despite additional educational interventions. Therapeutic education allows families in precarious situations to acquire, during the initial hospitalization, knowledge that meets the security objectives and is adapted to the care of their child. However, we have noticed that it can be difficult for some families to apply this knowledge when they are back in their home.

Thus, we are planning to set up a coordinated intervention by a pediatric nurse at the child's home to support the parents in the implementation of the theoretical knowledge acquired at the hospital.

Three home visits will be set up by a nurse during the first six months of the discovery of diabetes in the child. These visits will be organized during the first, fourth and sixth months after the discovery of diabetes and last about 2 hours each time. An additional visit may be set up according to the needs of families. The HbA1C measured 12 months after the diabetes diagnosis will be compared to the HbA1C obtained in an historical cohort that did not receive at-home therapeutic education.

ELIGIBILITY:
For the prospective group (strategy under study):

* 1 to 16 years old
* Diagnosis of type 1 diabetes (T1D)
* EPICES score > 30 (if separated parents, highest score)
* Hospitalized at the discovery of T1D in the pediatric diabetology unit of Bordeaux University Hospital
* Parents affiliated to social security
* Living in Gironde
* Consent of the parents or the holders of parental authority for the participation of their child
* Assent of the child

For the retrospective group (classic strategy):

* 1 to 16 years old at diabetes diagnosis
* Diagnosis of type 1 diabetes (T1D) from 1 January 2017 until the start of the study inclusion period
* EPICES score > 30 (if separated parents, highest score)
* Hospitalized to the discovery of T1D and followed by the pediatric diabetology unit of Bordeaux University Hospital
* Parents affiliated to social security
* Living in Gironde
* For patients who are minor at the time of the study: whose parents or holders of the parental authority have received an individual information and are not opposed to the use of their data (EPICES score and their child's clinical data).

For minors who became adults at the time of the study: having received individual information and are not opposed to the use of the data necessary for the study (EPICES score and their clinical data).

Exclusion criteria:

For the prospective group (strategy under study):

* Absence of the therapeutic education nurse during the child's hospitalization
* Child and/or family who do not speak French
* Family benefiting from the PASS
* Intention of leaving the Gironde department in the first six months of the study
* T1D with associated chronic pathological conditions other than hypothyroidism and celiac disease

For the retrospective group (classic strategy):

* Child and/or family who do not speak French
* Family benefiting from the PASS
* T1D with associated chronic pathological conditions other than hypothyroidism and celiac disease

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 29 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Measurement of HbA1c (%) one year after the discovery of diabetes. | 12 months after the diabetes diagnosis
  The Glycated hemoglobin (HbA1C) measured 12 months after the diabetes diagnosis

SECONDARY OUTCOMES:
Number of visits actually carried out in the interventional arm | 12 months after the diabetes diagnosis
  3 visits are planned but an additional visit may be set up according to the needs of families.
  It is also possible that some visits cannot take place. The number of visits actually made will therefore be recorded.
Evaluation of the satisfaction with the intervention of the children and parents | 12 months after the diabetes diagnosis
  Evaluation of the satisfaction with the intervention of the children and parents, measured with a standard visual analogue scale at the end of the intervention of the pediatric nurse
Evaluation of the satisfaction with the intervention of the pediatric endocrinology department's caregivers | 12 months after the diabetes diagnosis
  Evaluation of the satisfaction of the pediatric endocrinology department's caregivers (pediatric diabetologists, nurses, dieticians) with the intervention, measured with a standard visual analogue scale at the end of the intervention of the pediatric nurse
Evaluation of the satisfaction with the intervention of the external partners | 12 months after the diabetes diagnosis
  Evaluation of the satisfaction of the external partners (doctor or pediatrician, providers) with the intervention, measured with a standard visual analogue scale at the end of the intervention of the pediatric nurse
Unscheduled hospital visits in the context of T1D | Through study completion, 12 months after the diabetes diagnosis
  Number of emergency visits and hospitalizations
Percentage of time spent in the target for patients with Freestyle sensor | during the last month of the study, between 11 and 12 months after the diabetes diagnostic
  Percentage of time spent in the target (subcutaneous glucose measurement between 70 and 180 mg/dl) during the last month of the study for patients with Freestyle sensor
Percentage of time spent wearing the sensor for patients with Freestyle sensor | during the last month of the study, between 11 and 12 months after the diabetes diagnostic
  Percentage of time spent wearing the sensor during the last month of the study for patients with Freestyle sensor

CONTACTS AND LOCATIONS:
Overall Officials: Magali GIMENEZ, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Chu Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No